CLINICAL TRIAL: NCT01610921
Title: Determining the Optimal Dry Powder Adenosine Provocation Test to Assess Small Airways Disease
Brief Title: Determining the Optimal Adenosine Provocation Test
Acronym: impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, E. van der Wiel, E. van der Wiel, MD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL 37702.042.12
Record Dates: First submitted 2012-05-22; First posted 2012-06-04 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: asthma; small airways disease; inflammation; provocation; adenosine
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- bronchial provocationtest (Experimental): Provocation tests with adenosine dry powder and nebulized AMP (adenosine-5'monophosphate). The AMP provocation test is a standard test and consists of 14 doubling concentrations in a range of 0.04mg/ml to 320mg/ml. The aerosols will be inhaled during tidal breathing for 2 minutes. The dry powder adenosine also consists of 14 doubling steps with doses in a range of 0.01mg to 20mg.
  Interventions: Other: Bronchial provocation test

INTERVENTIONS:
Other: Bronchial provocation test — Provocation tests with adenosine dry powder and nebulized AMP (adenosine-5'monophosphate). The AMP provocation test is a standard test and consists of 14 doubling concentrations in a range of 0.04mg/ml to 320mg/ml. The aerosols will be inhaled during tidal breathing for 2 minutes. The dry powder adenosine also consists of 14 doubling steps with doses in a range of 0.01mg to 20mg.
  Other Names: bronchial challenge test; AMP test; adenosine bronchial provocation

SUMMARY:
Asthma is a frequently occurring inflammatory lung disease that affects the whole bronchial tree including the small airways (<2mm). Since the introduction of the solution hydrofluoroalkane (HFA) technology it is possible to generate medication with small particles of approximately 1-2 μm, and therefore to reach the small airways. However, at this moment the investigators have no reliable instruments to identify the asthmatic subjects who particularly benefit from treatment with inhaled small particles. Recently the investigators research group investigated whether provocation with small and large particles AMP is able to identify responders and non-responders to treatment with small and large particles of inhaled corticosteroids. This provocation technique gave promising results but needs further optimization.

The aim of this study is to determine the optimal particle size of dry powder adenosine to assess small airway involvement in asthma. Secondary, to provide insight in the associations between the standard test, executed with nebulized AMP, and the new test, executed with dry powder Adenosine.

DETAILED DESCRIPTION:
This is a cross-over study. The study population consists of 10 non-smoking asthma patients in the age of 18-65 years who have a PC20 metacholine value ≤4.9mg/ml.

Participating subjects perform 6 provocation tests in randomized order: one test with nebulized methacholine, one test with nebulized AMP, four times dry powder adenosine provocation test. (small particles with inhaled with a slow flow, small particles inhaled with a fast flow, large particles inhaled with a slow flow, large particles inhaled with a fast flow)

ELIGIBILITY:
Inclusion Criteria:

* A doctor's diagnosis of asthma
* Age: 18-65 years
* PC20 AMP < 320 mg/ml
* Non-smoker
* Steroid naive or steroids have been stopped 4 weeks before entry into the baseline period

Exclusion Criteria:

* Recent exacerbation asthma (<2 months) or upper respiration tract infection (<2 weeks)
* Severe airway obstruction at baseline, FEV1pred< 50% or < 1.2L
* Diagnosis of COPD or any other pulmonary disease that could influence the study results as judged by the investigator
* Pregnancy or lactating women. (i.e. women of childbearing potential who do not use adequate anticonception as judged by the investigator).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The small airway reaction to provocation with adenosine, reflected by the IOS parameter R5-R20 | Small airway reaction is measured during each provocation test. The Visits will take place in a period of 6 weeks.
  The R5-R20 is measured with the IOS. This a method to determine the resistance of the small airways. The R5-R20 is measured during each provocation test after each provocative step.

SECONDARY OUTCOMES:
The total airway reaction to provocation with adenosine, reflected by the decline in FEV1 (PD20/ PC20 values) | Lung function is measured during each provocation test. All visits take place in a period of 6 weeks.
  We want to compare the different PD20/PC20 values of the three dry powder adenosine provocation test and with the nebulized AMP provocation test. The lung function is measured after each provocative step to determine the point of 20% decline in FEV1. The provocation test is ended after the last step or is ended prematurely when there is a 20% fall of FEV1 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nick ten Hacken, MD, Phd, Study Chair — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - University Medical Center Groningen, Groningen